CLINICAL TRIAL: NCT04345536
Title: Prospective Quality Register of Patients With Confirmed Covid-19 at Oslo University Hospital
Acronym: CovidRegOUH
Status: Completed | Type: Observational
Sponsor: Oslo University Hospital (Other)
Responsible Party: Principal Investigator, Aleksander Rygh Holten, MD, Oslo University Hospital
Other Study IDs: CovidRegOUH
Record Dates: First submitted 2020-04-05; First posted 2020-04-14 (Actual); Last update posted 2023-11-14 (Actual); Status verified 2023-11

CONDITIONS: COVID-19
MeSH Terms: conditions — COVID-19

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Year
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Patients hospitalized with confirmed Covid-19: All patients hospitalized with confirmed Covid-19

SUMMARY:
Covid-19 is a recently emerging infectious disease with a very large impact on health care world-wide. The disease is still poorly described. It is an urgent need for better clinical characteristics. A prospective, quality register is therefore established for increasing the knowledge about the disease, the covid patients and the prognosis.

DETAILED DESCRIPTION:
All patient hospitalized at Oslo University Hospital, Ullevål, is prospectively registered in the approved quality register. Background, clinical and paraclinical data is harvested and registered, as well as treatment and mortality.

ELIGIBILITY:
Inclusion Criteria:

* Confirmed covid-19
* hospitalized

Exclusion Criteria:

* None

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Hospitalized patients in a secondary and tertiary care University Hospital.
Sampling Method: Probability Sample
Enrollment: 2519 (Actual)
Dates: Start 2020-03-15 (Actual); Primary Completion 2022-01-01 (Actual); Study Completion 2023-11-01 (Actual)

PRIMARY OUTCOMES:
Mortality | 3 month
  Mortality in hospitalized covid patients
Severe disease | 2 weeks
  Number of patients with severe disease

CONTACTS AND LOCATIONS:
Overall Officials: Kristian Tonby, MD, Study Director — Oslo University Hospital
Locations (1):
- Oslo University Hospital, Oslo, Norway

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Holten AR, Nore KG, Tveiten CEVWK, Olasveengen TM, Tonby K. Predicting severe COVID-19 in the Emergency Department. Resusc Plus. 2020 Dec;4:100042. doi: 10.1016/j.resplu.2020.100042. Epub 2020 Oct 21. PMID 33403367